CLINICAL TRIAL: NCT04783311
Title: A Phase 1/2 Dose-exploration, Randomized, Observer-blind, Placebo-controlled Study to Determine Safety, Tolerance and Immunogenicity of EuCorVac-19, a Recombinant Protein Vaccine, for the Prevention of COVID-19 in Healthy Adults
Brief Title: Safety, Tolerance and Immunogenicity of EuCorVac-19 for the Prevention of COVID-19 in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EuSNAP_COV101
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1 - EuCorVac-19 Low dose group (Experimental): Healthy adults received two intramuscular doses (0.5mL per dose) with 3-week interval
  Interventions: Biological: EuCorVac-19; Other: Normal Saline
- Phase 1 - EuCorVac-19 High dose group (Experimental): Healthy adults received two intramuscular doses (0.5mL per dose) with 3-week interval
  Interventions: Biological: EuCorVac-19; Other: Normal Saline
- Phase 2 - EuCorVac-19 Low dose group (Experimental): Healthy adults received two intramuscular doses (0.5mL per dose) with 3-week interval
  Interventions: Biological: EuCorVac-19
- Phase 2 - EuCorVac-19 High dose group (Experimental): Healthy adults received two intramuscular doses (0.5mL per dose) with 3-week interval
  Interventions: Biological: EuCorVac-19
- Phase 2 - Placebo comparator group (Active Comparator): Healthy adults received two intramuscular doses (0.5mL per dose) with 3-week interval
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: EuCorVac-19 — Two intramuscular doses (0.5mL per dose) at 3-week interval
  Arms: Phase 1 - EuCorVac-19 High dose group; Phase 1 - EuCorVac-19 Low dose group; Phase 2 - EuCorVac-19 High dose group; Phase 2 - EuCorVac-19 Low dose group
Other: Normal Saline — Two intramuscular doses (0.5mL per dose) at 3-week interval
  Arms: Phase 1 - EuCorVac-19 High dose group; Phase 1 - EuCorVac-19 Low dose group; Phase 2 - Placebo comparator group

SUMMARY:
Phase I/II study to determine safety, tolerance and immunogenicity of EuCorVac-19, a recombinant protein vaccine, for the prevention of COVID-19 in healthy adults

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who voluntarily decide to participate in this study and provide written informed consent

   * Healthy male and female adult at the age of 19 to 50 years (Part A)
   * Healthy male and female adult at the age of 19 to 75 years (Part B)
2. Individuals who are available for all visit procedures including telephone visits during the study period

Exclusion Criteria:

1. COVID-19 positive based on RT-PCR using upper respiratory tract or lower respiratory tract sampling or COVID-19 antibody positive
2. History of SARS-CoV, MERS-CoV or SARS-CoV-2 infection
3. History of vaccination against SARS-CoV, MERS-CoV or SARS-CoV-2
4. Immune system disorders including immunodeficiency disease
5. Clinically significant abnormalities in clinical laboratory test, ECGs and chest X-ray during screening in the opinion of the investigator
6. Fever within 3 days prior to screening or serious acute or chronic infection within 7 days prior to screening requiring systemic antibiotics or antivirals
7. Evidence or history of serious acute, chronic, or progressive disease which, in the opinion of the investigator, makes the individual ineligible for the study
8. History of severe allergic reactions or severe hypersensitivity reactions to the IP or any of its components
9. History of therapy that might affect immunity: treatment with immunosuppresants or immune modifying drugs, anticancer therapy, or radiotherapy within 3 months prior to screening
10. Women of childbearing potential who do not agree to use medically allowed methods of contraception or to be heterosexually inactive until 60 days after the last dose of the IP
11. Pregnant or breastfeeding woman
12. Treatment with other IPs within 6 months prior to participation in this study
13. Other reasons including medical reasons based on which the individual is considered to be ineligible for this study in the opinion of the investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Immediate AEs | within 30 minutes after each IP dosing
Solicited local and systemic AEs | for 7 days after each IP dosing
Unsolicited AEs | within 28 days after the last IP dosing
SAEs | within 52 weeks after the last IP dosing
AESIs | within 52 weeks after the last IP dosing

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Eunpyeong St.Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lovell JF, Baik YO, Choi SK, Lee C, Lee JY, Miura K, Huang WC, Park YS, Woo SJ, Seo SH, Kim JO, Song M, Kim CJ, Choi JK, Kim J, Choo EJ, Choi JH. Interim analysis from a phase 2 randomized trial of EuCorVac-19: a recombinant protein SARS-CoV-2 RBD nanoliposome vaccine. BMC Med. 2022 Nov 30;20(1):462. doi: 10.1186/s12916-022-02661-1. PMID 36447243
- [Derived] Sia ZR, He X, Zhang A, Ang JC, Shao S, Seffouh A, Huang WC, D'Agostino MR, Teimouri Dereshgi A, Suryaprakash S, Ortega J, Andersen H, Miller MS, Davidson BA, Lovell JF. A liposome-displayed hemagglutinin vaccine platform protects mice and ferrets from heterologous influenza virus challenge. Proc Natl Acad Sci U S A. 2021 Jun 1;118(22):e2025759118. doi: 10.1073/pnas.2025759118. PMID 34050027